CLINICAL TRIAL: NCT03543735
Title: A Targeted, Real-Time, Technology-Supported Intervention for Patients With Alcohol Use Disorder on Disulfiram
Acronym: Wisepill+SMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1804-001
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Drinking, Alcohol
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Disulfiram usage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wisepill+SMS (Experimental)
  Interventions: Behavioral: Wisepill+SMS
- Wisepill-only (Active Comparator)
  Interventions: Other: Wisepill-only
- Disulfiram-only (No Intervention)

INTERVENTIONS:
Behavioral: Wisepill+SMS — This will include: 1) an in-person Wisepill orientation session to introduce the pillbox and generate relapse prevention messages that can be later delivered during non-adherent windows; 2) use of the Wisepill device during the intensive treatment program and after discharge; and 3) three forms of tailored SMS messages paired with Wisepill device use: a) supportive messages with medication compliance, b) reminder messages for early non-adherence (e.g., 1 hour late) and c) relapse-prevention messages after longer periods of non-adherence (e.g., several hours).
  Arms: Wisepill+SMS
Other: Wisepill-only — This will include: 1) an in-person Wisepill orientation session to introduce the pillbox; 2) use of the Wisepill during the intensive treatment program and after discharge.
  Arms: Wisepill-only

SUMMARY:
Alcohol use disorders (AUDs) are a costly and burdensome health concern, affecting over 15 million adults each year in the United States. Several FDA-approved medication-assisted therapies (MATs) are used for the treatment of AUD, with disulfiram (Antabuse) the oldest and one of the most common. Disulfiram acts as a "psychological deterrent" and causes physiological reactions when taken with alcohol. Despite demonstrated efficacy for decreasing relapse, disulfiram is underutilized: efficacy is best demonstrated under monitoring or supervision, creating a barrier for use. Additionally, disulfiram adherence rates are low. The most common reason for non-adherence is that an individual is contemplating or planning a relapse, which typically occurs within 50 hours. Thus, disulfiram non-adherence can be a marker for relapse, providing a very short window for intervention. Technological advances now allow for electronic medication monitoring: devices are designed to objectively track adherence. The Wisepill device is an electronic medication monitoring system that pairs real-time monitoring with a triggered text message (SMS) when doses are late. The Wisepill device plus medication reminder SMS messages are associated with increased adherence to antiretroviral or diabetic therapy. Though the capability exists, potentially therapeutic SMS messages paired with Wisepill objective monitoring have yet to tested in any population. Indeed, previous research suggests that supportive and relapse prevention/coping skills SMS message interventions are effective in reducing alcohol use. Thus, given that disulfram non-adherence can signify a critical clinical concern (i.e., impending relapse), the delivery of a tailored, relapse prevention-focused, just-in-time SMS soon after disulfiram discontinuation could have a significant impact on AUD treatment outcomes. The investigators propose to develop an intervention capitalizing on the Wisepill technology to pair real-time medication monitoring with tailored (a) real-time triggered reminders, (b) real-time abstinence support, and (c) relapse prevention SMS texts for individuals with AUD being treated with disulfram.

The investigators propose to develop a 12-week Wisepill+SMS intervention for individuals in alcohol treatment on disulfiram. This will include: 1) an in-person Wisepill orientation session to introduce the device and generate tailored relapse prevention messages; 2) use of the Wisepill device during the intensive treatment program and after discharge; 3) tailored SMS messages paired with use of the Wisepill device: a) supportive messages with medication compliance, b) reminder messages for early non-adherence (e.g., 1 hour late) and c) relapse-prevention messages after longer periods of non-adherence (e.g., several hours). The goal of this application is to develop the Wisepill+SMS intervention with the aid of focus groups (n=20), then test the Wisepill+SMS intervention in a RCT (n=75) comparing Wisepill+SMS to Wisepill only (i.e., no SMS) and disulfiram only (i.e., no Wisepill, no SMS). The Wisepill device, and its associated real-time monitoring and messaging systems, are relatively low-cost, easy to program, and can deliver an intervention that would reduce barriers to care.

DETAILED DESCRIPTION:
Excessive alcohol use is associated with a host of economic and health problems, with an estimated annual burden of over $249 billion. One-third of the population will meet diagnostic criteria for alcohol use disorder (AUD) in their lifetime. Among those who become abstinent, relapse rates are high, particularly in the first 90 days of sobriety. Pharmacotherapy continues to be an effective treatment approach. Several FDA-approved medication-assisted therapies are used, commonly disulfiram (Antabuse) 5. Disulfiram acts as a "psychological deterrent" and causes physiological reactions when taken with alcohol. Despite demonstrated efficacy for decreasing relapse, disulfiram is underutilized, primarily because of the supervision and monitoring required for its most efficacious use. In addition, disulfiram adherence rates are low. Reasons for non-adherence may be non-deliberate (i.e., forgetfulness), but often are deliberate (i.e., contemplating or planning a relapse to alcohol use). Indeed, individuals who discontinue disulfiram relapse approximately 50 hours after a missed dose 4. Thus, disulfiram discontinuation may be a proxy for a return to drinking. Identifying this window before relapse, through medication monitoring and implementing a just-in-time intervention, may reduce risk of relapse.

Previous methods used to monitor adherence have been subject to self-report bias, have been constrained by the need for observer reports, have measured prescription refills as a proxy for adherence, or have relied on participant attendance at later assessment sessions to collect data. Technological advances now offer the opportunity to objectively measure adherence in real time through opening of the medication bottle. The Wisepill device is an electronic medication event monitoring systems that can pair real-time monitoring with a triggered text message (Short Message Service; SMS) when doses are late. Studies utilizing Wisepill plus medication reminder SMS messages find increased adherence to antiretroviral or diabetic therapy. Though the capability exists, potentially therapeutic SMS messages paired with Wisepill objective monitoring have yet to tested. Given that disulfram non-adherence can signify a potentially critical clinical concern (i.e., impending relapse), the delivery of a tailored, relapse prevention-focused, just-in-time message soon after a disulfiram dose has been missed could have a significant impact on AUD treatment outcomes. Indeed, previous research suggests that supportive and relapse prevention/coping skills SMS message interventions are effective in reducing rates of alcohol use. The investigators propose to develop an intervention capitalizing on the Wisepill technology to pair real-time medication monitoring with tailored (a) real-time triggered reminders, (b) real-time abstinence support, and (c) relapse prevention SMS texts for individuals with AUD being treated with disulfram.

PRIMARY AIMS

1. To develop a 12-week Wisepill+SMS intervention for individuals in intensive outpatient alcohol treatment who are prescribed disulfram. This will include: 1) an in-person Wisepill orientation session to introduce the device and generate relapse prevention messages that can be later delivered during non-adherent windows; 2) use of the Wisepill device during the intensive treatment program and after discharge; and 3) three forms of tailored SMS messages paired with Wisepill device use: a) supportive messages with medication compliance, b) reminder messages for early non-adherence (e.g., 1 hour late) and c) relapse-prevention messages after longer periods of non-adherence (e.g., several hours).

1a. The investigators will conduct 4 focus groups (total n=20) with patients previously (2 groups) and currently (2 groups) prescribed disulfram to help identify barriers to the Wisepill+SMS intervention, inform the types of SMS messages to be delivered, and determine strengths and limitations of the proposed intervention.

1b. The investigators will modify and finalize the Wisepill+SMS intervention, based on data from focus groups, as well as barriers limiting its utility.

2. To conduct a preliminary RCT with 75 individuals with AUD utilizing disulfiram in early recovery, comparing (a) Wisepill+SMS intervention, (b) monitoring by Wisepill only (i.e., no SMS texts delivered), and (c) disulfiram use only (i.e., no Wisepill). The investigators hypothesize: 2a. Relative to the Wisepill-only and disulfiram-only conditions, the Wisepill+SMS condition will demonstrate improved outcomes with regard to the primary outcome of interest (i.e., alcohol use), specifically greater percent days abstinent at end of intervention (3-months) and at 6-month follow-up.

2b. Relative to the Wisepill-only and disulfiram-only conditions, the Wisepill+SMS condition will result in greater adherence to medication, increased coping, increased self-efficacy, and increased perceived social support.

2c. The investigators hypothesize that these mechanisms (i.e., medication adherence, coping strategy utilization, abstinence self-efficacy, and perceived social support) will be significantly associated with alcohol outcomes.

The investigators anticipate that this project will lead to the development of a well-specified, novel, technology-supported medication adherence/relapse prevention intervention for individuals with AUD utilizing disulfiram in early recovery that can be subsequently tested in a future fully-powered randomized controlled treatment trial.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years of age
* meet DSM-5 criteria for an AUD, as assessed by the SCID-P,
* prescribed disulfiram while in the Alcohol and Drug Partial Hospital Program (i.e., while also meeting psychiatrist criteria for a disulfiram protocol)
* are currently enrolled in ADP
* has access to a phone capable of receiving SMS and access to email.

Exclusion Criteria:

* current DSM-5 diagnosis moderate/severe substance use disorder
* a history of psychotic disorder or current psychotic symptoms
* current suicidality or homicidality
* current use of an alcohol treatment medication other than disulfiram.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Timeline Followback (TLFB) for alcohol use | 6 months
  Alcohol use, yes/no for last 90 days or since last assessment
Alcohol breath analysis | 6 months
  Breathalyser
PEth blood alcohol testing | 6 months
  Biological measure of alcohol use
Wisepill adherence counts | 6 months
  Record of use of Wisepill pillbox
Zenalyser Antabuse breath compliance test | 6 months
  Test of disulfiram (Antabuse) metabolites
Self-reported medication adherence | 6 months
  Self-reported use of disulfiram

SECONDARY OUTCOMES:
Multidimensional Scale of Perceived Social Support | 6 months
  Perceived social support, 12 items (measured 1-7, total=12-84, higher=more perceived support)
Alcohol Abstinence Self-Efficacy Scale | 6 months
  Belief in ability to abstain from alcohol, 40 items (measured 0-4, total=0-160, higher=more self-efficacy)
Brief COPE | 6 months
  Coping skills and strategies, 28 items (measured 1-4) and 14 subscales. Subscale scores will be used (range in scores = 2-8, higher=more use of coping strategy)

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No